CLINICAL TRIAL: NCT02058472
Title: An Open Label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetic/Pharmacodynamic Characteristics and Safety Following Administration of G3041 and SEVIKAR® Tablet in Healthy Adult Volunteers
Brief Title: Pharmacokinetic/Pharmacodynamic & Safety Study of G3041 and SEVIKAR® Tablet in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G3041_BE_I
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G3041 (Experimental): Amlodipine orotate 10mg/Olmesartan medoxomil 40mg
  Interventions: Drug: G3041; Drug: SEVIKAR®
- SEVIKAR® (Active Comparator): Amlodipine besylate 10mg/Olmesartan medoxomil 40mg
  Interventions: Drug: G3041; Drug: SEVIKAR®

INTERVENTIONS:
Drug: G3041
Drug: SEVIKAR®

SUMMARY:
Study Design : randomized, open label, single-dose, 2-way cross-over design

Phase : Phase I

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between the ages of 19 to 55 years old
* 19 ≤ BMI ≤ 27
* having neither congenital/chronic diseases nor pathological symptoms/findings as results of medical examination
* doctor determines to be suitable as subjects within 4 weeks ago before administration

Exclusion Criteria:

* Hypersensitivity(or history of hypersensitivity) to amlodipine and olmesartan
* Exceed 1.5 times of the upper limit of the reference range of AST, ALT, total bilirubin, γ-GT
* Excessive drinking(exceed alcohol 140g/week)
* Excessive caffeine(exceed 4cups/day) and grape fruit/orange juice(exceed 1cup/day)
* Smoking over 10 cigarettes per day

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
AUClast, Cmax | Blood gathering point : 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 7h, 8h, 12h, 24h, 48h, 72h

SECONDARY OUTCOMES:
tmax, t1/2, AUCinf, CL/F, Vz/F | Blood gathering point : 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 7h, 8h, 12h, 24h, 48h, 72h
ΔAUEC24, ΔEmax, tEmax | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 24h, 48h, 72h

CONTACTS AND LOCATIONS:
Overall Officials: JW Ko, MD, PhD, Principal Investigator — Samsung Medical Center